CLINICAL TRIAL: NCT02111174
Title: A Pilot Randomized Sham-Controlled Trial of MC5-A Calmare Therapy (Scrambler Therapy) in the Treatment of Chronic Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Scrambler Therapy in the Treatment of Chronic Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: J1384; J1384 (Other: SKCCC at Johns Hopkins); NA_00086429 (Other: JHMIRB)
Record Dates: First submitted 2014-03-23; First posted 2014-04-11 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Neuropathy
Keywords: Neuropathy; Peripheral neuropathy; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scrambler Therapy (Experimental): The device is a cutaneous electrical stimulator that uses electrodes placed on the skin similar to an electrocardiogram (EKG) machine, feeling similar to a tingling or bee-sting like sensation during the therapy. The electrodes are placed in areas thought to help relieve pain associated with chemotherapy-induced peripheral neuropathy.
  Interventions: Device: Scrambler Therapy
- Sham Therapy (Sham Comparator): The device is a cutaneous electrical stimulator that uses electrodes placed on the skin similar to an electrocardiogram (EKG) machine, feeling similar to a tingling or bee-sting like sensation during the therapy. The electrodes are placed in areas not thought to help relieve pain associated with chemotherapy-induced peripheral neuropathy.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Scrambler Therapy
  Other Names: MC5-A Calmare Therapy; Scrambler ST 5 TENS Device
  Arms: Scrambler Therapy
Device: Sham Therapy
  Arms: Sham Therapy

SUMMARY:
The purpose of this study is to see if Scrambler Therapy with the Calmare MC5-A machine will relieve chemotherapy induced peripheral neuropathy (CIPN).

Scrambler Therapy is a method of pain relief given with common electrocardiography (ECG) skin electrodes. The electrodes are placed on the body in pairs, and the Scrambler Therapy machine directs electrical signals across the field to simulate non-pain information.

Based on other studies, we think that we relieve pain with the Scrambler therapy device, but it has not been tested in a setting such as this one. This means that some of the pain relief could be due to placebo effect, or the CIPN pain going away on its own. In this study we want to compare the Scrambler Therapy with the sham therapy (the therapy that does not use the electrical signals). We hope that this study will help us determine if the Scrambler device really helps patients with CIPN.

Cancer patients with chronic, chemotherapy-related pain of 4 or more (on a 0-10 scale) for at least 3 months may be eligible to join this study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years of age or older with cancer
* English speakers
* Lower extremity CIPN neuropathy: Received neurotoxic chemotherapy (including taxanes-such as paclitaxel or docetaxel, or platinum-based compounds such as carboplatin or cis-platinum or oxaliplatin, or vinca alkaloids such as vincristine, vinblastine, or vinorelbine, or proteosome inhibitors such as bortezimib).
* Pain or symptoms of lower extremity peripheral neuropathy of >3 month's duration attributed to chemotherapy-induced peripheral neuropathy
* An average daily pain rating of > 4 out of 10
* Life expectancy >3 months
* ECOG Performance Status 0, 1, 2, or 3
* Patient understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form

Exclusion Criteria:

* Any of the following: pregnant women, nursing women, women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, abstinence, etc.).
* Use of an investigational agent for pain control concurrently or within the past 30 days
* History of an allergic reaction or previous intolerance to transcutaneous electronic nerve stimulation
* Patients with implantable drug delivery systems, e.g. Medtronic Synchromed
* Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, cochlear implants, aneurysm clips, vena cava clips and skull plates. (Metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed)
* Patients with a history of myocardial infarction or ischemic heart disease within the past six months
* Patients with history of epilepsy, brain damage, or symptomatic brain metastases
* Prior celiac plexus block, or other neurolytic pain control treatment
* Other identified causes of painful parasthesias existing prior to chemotherapy (e.g., radiation or malignant plexopathy, lumbar or cervical radiculopathy, pre-existing peripheral neuropathy of another etiology: e.g., carpal tunnel syndrome, B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy, etc.) that might be responsible for the patient's current neuropathic symptoms
* Skin conditions such as open sores that would prevent proper application of the electrodes
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study
* Currently receiving anti-convulsants (such as gabapentinoids, e.g. gabapentin (Neurontin) or pregabalin (Lyrica). Because of data that support that patients do not do as well when on gabapentin or pregabalin, all patients on these medications will be weaned off them prior to study initiation. The study team will provide instructions on how to do this

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Smith, MD, FACP, Principal Investigator — SKCCC at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cathcart-Rake EJ, Hilliker DR, Loprinzi CL. Chemotherapy-induced neuropathy: Central resolution of a peripherally perceived problem? Cancer. 2017 Jun 1;123(11):1898-1900. doi: 10.1002/cncr.30650. Epub 2017 Mar 3. No abstract available. PMID 28257145

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was consented and enrolled for training purposes only with the scrambler machine. This participant was not randomized into an arm and was not used in analysis.
Groups:
- Scrambler Therapy: The device is a cutaneous electrical stimulator that uses electrodes placed on the skin similar to an electrocardiogram (EKG) machine, feeling similar to a tingling or bee-sting like sensation during the therapy. The electrodes are placed in areas thought to help relieve pain associated with chemotherapy-induced peripheral neuropathy.
  Scrambler Therapy
- Sham Therapy: The device is a cutaneous electrical stimulator that uses electrodes placed on the skin similar to an electrocardiogram (EKG) machine, feeling similar to a tingling or bee-sting like sensation during the therapy. The electrodes are placed in areas not thought to help relieve pain associated with chemotherapy-induced peripheral neuropathy.
  Sham Therapy
Period: Treatment and Primary Outcome
Arm/Group | Scrambler Therapy | Sham Therapy
Started | 18 | 18
Completed | 15 | 16
Not Completed | 3 | 2
Not completed — Ineligible (not used in analysis) | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Period: Secondary Outcomes (2 and 3 Month f/u)
Arm/Group | Scrambler Therapy | Sham Therapy
Started | 15 | 16
2 Month Follow up Complete | 8 | 11
Completed | 7 | 9
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 8 | 6
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant in the scrambler therapy arm was determined to be ineligible retrospectively and they did not complete treatment on the study, therefore they were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Scrambler Therapy | Sham Therapy | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.71 (8.88) | 58.94 (9.31) | 59.31 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Pain Score [Mean (Standard Deviation); unit: units on a scale] — Change in pain as measured by the Modified Brief Pain Index (BPI), question #3. The BPI short form is a pain assessment tool used with cancer patients to measure both severity of pain and interference caused by pain on 0-10 scales with higher scores indicating more pain.
  units on a scale | 6.29 (1.9) | 6.83 (1.62) | 6.57 (1.75)
Using opioids at baseline or during treatment [Count of Participants; unit: Participants] — This will be assessed by concomitant medication review by a study team member during the 10 days of treatment. Follow-up was assessed as participant self-report over the last 10 days; all opiates were further tabulated using a morphine oral dose equivalents table to allow better comparison between patients and arms.
  Participants | 5 | 3 | 8
Using neuroleptics at baseline or during treatment [Count of Participants; unit: Participants] — This will be assessed by concomitant medication review by a study team member during the 10 days of treatment. Follow-up was assessed as participant self-report over the last 10 days; all opiates were further tabulated using a morphine oral dose equivalents table to allow better comparison between patients and arms.
  Participants | 3 | 4 | 7
Sensory subscale score at baseline [Mean (Standard Deviation); unit: units on a scale] — This was assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CIPN20, a CIPN-specific questionnaire which includes two scales assessing sensory and motor symptoms and functioning with each question measured on a 0-3 scale. For sensory there are 9 questions with a total score range from 0-27 with higher scores indicating more bothersome symptoms.
  units on a scale | 13.47 (5.73) | 15.83 (4.49) | 14.69 (5.19)
Motor subscale score at baseline [Mean (Standard Deviation); unit: units on a scale] — This will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CIPN20, a CIPN-specific questionnaire which includes two scales assessing sensory and motor symptoms and functioning with each question measured on a 0-3 scale. For motor there are 8 questions with a total score range from 0-24 with higher scores indicating more bothersome symptoms.
  units on a scale | 10.53 (5.21) | 11.83 (5.09) | 11.2 (5.12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain as Measured by the Modified Brief Pain Index at 28 Days
Description: To determine the change in pain from day 0 to day 28 (as measured by the Modified Brief Pain Index (BPI), question #3) with scrambler therapy in patients with chemotherapy induced peripheral neuropathy and pain (CIPN). The BPI short form is a pain assessment tool used with cancer patients to measure both severity of pain and interference caused by pain on 0-10 scales with higher scores indicating more pain. A negative score for the change in pain indicates improvement.
Time Frame: Change from baseline to 28 days
Population: Data was analyzed from 17/18 participants in Arm 1 since one was deemed ineligible in retrospect.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 17 | 18
units on a scale | -0.5 (1.2) | -1.06 (2.32)

2. Secondary Outcome: Change in Pain at 2 Months as Measured by the Modified Brief Pain Index
Description: To determine the change in pain from day 0 to 2 months (as measured by the Modified Brief Pain Index (BPI), question #3) with scrambler therapy in patients with chemotherapy induced peripheral neuropathy and pain (CIPN). The BPI short form is a pain assessment tool used with cancer patients to measure both severity of pain and interference caused by pain on 0-10 scales with higher scores indicating more pain. A negative score for the change in pain indicates improvement.
Time Frame: Change from baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 15 | 16
units on a scale | -0.31 (0.8) | -0.25 (0.92)

3. Secondary Outcome: Change in Pain at 3 Months as Measured by the Modified Brief Pain Index
Description: To determine the change in pain from day 0 to 3 months (as measured by the Modified Brief Pain Index (BPI), question #3) with scrambler therapy in patients with chemotherapy induced peripheral neuropathy and pain (CIPN). The BPI short form is a pain assessment tool used with cancer patients to measure both severity of pain and interference caused by pain on 0-10 scales with higher scores indicating more pain. A negative score for the change in pain indicates improvement.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 15 | 16
units on a scale | -0.75 (1.78) | -0.44 (1.12)

4. Secondary Outcome: Changes in Patient Reported Sensory Outcomes at 28 Days
Description: This was assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CIPN20, a CIPN-specific questionnaire which includes two scales assessing sensory and motor symptoms and functioning with each question measured on a 0-3 scale. For sensory there are 9 questions with a total score range from 0-27 with higher scores indicating more bothersome symptoms. A negative change in score indicates improvement in symptoms.
Time Frame: Change from baseline to 28 days
Population: Data was analyzed from 17/18 participants in Arm 1 since one was deemed ineligible in retrospect.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 17 | 18
units on a scale | -4.76 (6.69) | -4.67 (6.66)

5. Secondary Outcome: Changes in Patient Reported Sensory Outcomes at 2 Months
Description: as for outcome 4
Time Frame: Change from baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 15 | 16
units on a scale | -8.94 (9.33) | -8.39 (8.37)

6. Secondary Outcome: Changes in Patient Reported Sensory Outcomes at 3 Months
Description: as for outcome 4
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 15 | 16
units on a scale | -9.62 (9.22) | -11.39 (7.84)

7. Secondary Outcome: Changes in Patient Reported Motor Outcomes at 28 Days
Description: This will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CIPN20, a CIPN-specific questionnaire which includes two scales assessing sensory and motor symptoms and functioning with each question measured on a 0-3 scale. For motor there are 8 questions with a total score range from 0-24 with higher scores indicating more bothersome symptoms. A negative change in score indicates improvement in symptoms.
Time Frame: Change from baseline to 28 days
Population: Data was analyzed from 17/18 participants in Arm 1 since one was deemed ineligible in retrospect.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 17 | 18
units on a scale | -2.97 (6.49) | -2.83 (6.35)

8. Secondary Outcome: Changes in Patient Reported Motor Outcomes at 2 Months
Description: as for outcome 7
Time Frame: Change from baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 15 | 16
units on a scale | -5.88 (7.27) | -5.67 (6.59)

9. Secondary Outcome: Changes in Patient Reported Motor Outcomes at 3 Months
Description: as for outcome 7
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 15 | 16
units on a scale | -6.62 (6.59) | -8.53 (7.28)

10. Secondary Outcome: Number of Patients Who Stopped Using Opioids at 28 Days
Description: This will be assessed by concomitant medication review by a study team member during the 10 days of treatment. Follow-up was assessed as participant self-report over the last 10 days; all opiates were further tabulated using a morphine oral dose equivalents table to allow better comparison between patients and arms.
Time Frame: 28 days post-intervention
Population: Data was analyzed from 17/18 participants in Arm 1 since one was deemed ineligible in retrospect.
Measure: Count of Participants; unit: Participants
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 17 | 18
Participants | 3 | 1

11. Secondary Outcome: Number of Patients Who Stopped Using Neuroleptics at 28 Days
Description: as for outcome 10
Time Frame: 28 days post-intervention
Population: Data was analyzed from 17/18 participants in Arm 1 since one was deemed ineligible in retrospect.
Measure: Count of Participants; unit: Participants
Arm/Group | Scrambler Therapy | Sham Therapy
Number analyzed (Participants) | 17 | 18
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 3 months after participants initiated treatment.
Description: AEs were self reported by participants as they occurred and collected between the time participants initiated treatment to the time they completed all treatment and follow up on the study at 3 months.
Arm/Group | Scrambler Therapy | Sham Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scrambler Therapy (N=18) | Sham Therapy (N=18)
Surgical and medical procedures - other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) — "Jolt" feeling and pain in left leg, transient from Scrambler Therapy with Calmare MC-5A device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02111174/Prot_SAP_000.pdf